CLINICAL TRIAL: NCT03014115
Title: EFFECTS OF DIFFERENT ARA FORMULATIONS OF INFANT FORMULA ON FATTY ACID STATUS, IMMUNE MARKERS AND INFECTION RATES IN INFANTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: SynteractHCR (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-1080
Record Dates: First submitted 2017-01-03; First posted 2017-01-09 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Healthy Infants
Keywords: arachidonic; docosahexaenoic acid; infant formula
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- combination ARA+ DHA (Active Comparator): combination 0.76% ARA+ 0.4% DHA in infant formula per day
  Interventions: Dietary Supplement: combination ARA + DHA
- DHA (Experimental): 0% ARA +0.4% DHA in infant formula per day
  Interventions: Dietary Supplement: DHA

INTERVENTIONS:
Dietary Supplement: combination ARA + DHA — combination ARA + DHA supplemented infant formula
  Other Names: infant formula
  Arms: combination ARA+ DHA
Dietary Supplement: DHA — DHA supplemented infant formula
  Other Names: infant formula
  Arms: DHA

SUMMARY:
The clinical trial will investigate the effect of different formulations of ARA + 0.4% DHA in infant formula on plasma fatty acid status in healthy 6 months old infants supplemented for 6 months. A 6-month follow on phase will provide additional efficacy (e.g. infection rates, immune markers) and safety information in these 12-18 month old infants.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, parallel-group study of 0% ARA +0.4% DHA or 0.76% ARA +0.4% DHA supplemented infant formula provided to 6 months old healthy infants for 6 months. Infants will have been breast-fed or formula-fed prior to enrollment. The difference in total plasma fatty acid ARA levels between the two groups at 6 months of supplementation will be measured. Parents will be asked about the infant's current daily diet (fatty acid intakes calculated via 24 hour recalls). All completed infants will be enrolled into a 6 month extension period (non-supplemented) to collect additional measures of efficacy (i.e. infections and illnesses, immune markers) and safety out to 18 months of age.

ELIGIBILITY:
Inclusion Criteria:

* singleton infants,
* parent of legal age to consent,
* willing to feed the child the assigned study formula for the treatment duration,
* parent agrees to scheduled blood draws

Exclusion Criteria:

* exclusively breastfed or formula-fed beyond 6 months,
* difficulty swallowing or other congenital malformation or metabolic anomaly,
* taking omega-3 (supplemented) foods,
* mother had gestational diabetes or is Type II diabetic,
* born at <37 weeks gestational age,
* participating in another study

Ages: 22 Weeks to 26 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2016-11; Primary Completion 2019-05 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
total plasma fatty acid ARA levels | 6 months of supplementation
  difference in total plasma fatty acid ARA levels between the two groups at 6 months of supplementation

SECONDARY OUTCOMES:
incidence of infections | 6 months of supplementation
  record number, type and duration of infections
weight gain | 6 months of supplementation
  differences between groups in weight gain (kg/d)
length gain | 6 months of supplementation
  differences between groups in length gain (cm/d)
head circumference | 6 months of supplementation
  differences between groups in head circumference (cm/d)
dietary intake of ARA | 6 months of supplementation
  24 hour recall questionnaire
plasma levels of immune markers | 6 months of supplementation
  cytokines and T cells levels in plasma will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Ascension Marcos, PhD, Principal Investigator — Instituto de Ciencia y Tecnología de Alimentos y Nutrición
Locations (2):
- Spain (2):
  - Centro de Salud Aravaca, Madrid
  - Centro Salud Arganda del Rey, Madrid

IPD SHARING:
Plan to Share IPD: No